CLINICAL TRIAL: NCT06202989
Title: Multiprofen-CC™ to Reduce Pain After Total Knee Arthroplasty: A Blinded Randomized Controlled Trial
Brief Title: Multiprofen-CC™ to Reduce Pain After Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: KAZM Pharmaceuticals Inc. (Industry)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-001
Record Dates: First submitted 2023-12-06; First posted 2024-01-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Postsurgical Pain
Keywords: Osteoarthritis, Knee; Arthroplasty, Replacement, Knee; Analgesics, Opioid
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: 2-arm parallel group randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All included patients, research personnel, healthcare providers and outcome assessors will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiprofen-CC™ (Experimental): Standard care pain medications and topical Multiprofen-CC™ (1g TID) for 6 weeks after surgery
  Interventions: Drug: Multiprofen-CC™ plus standard treatment
- Control (Placebo Comparator): Standard care pain medications and visually identical topical placebo (1g TID) for 6 weeks after surgery
  Interventions: Other: Placebo plus standard treatment

INTERVENTIONS:
Drug: Multiprofen-CC™ plus standard treatment — Multiprofen-CC™ [ketoprofen (10%), baclofen (5%), amitriptyline (2%), and lidocaine (5%)] Dose: 1.0g, 3 times per day for 6 weeks after surgery
  Arms: Multiprofen-CC™
Other: Placebo plus standard treatment — The placebo is the base cream with no medicinal ingredients to be applied 3 times per day for 6 weeks after surgery
  Other Names: Placebo
  Arms: Control

SUMMARY:
Total knee arthroplasty is a surgical treatment which involves replacing the damaged articular cartilage of the knee joint with an artificial prosthetic in end-stage knee osteoarthritis. Although total knee arthroplasties are mostly successful, approximately 1 in 5 patients are unsatisfied with their outcomes with 16-33% of patients of patients experiencing lasting pain following total knee arthroplasty.

Multiprofen-CC™ is a compounded topical analgesic currently available to healthcare professionals for prescription in patients experiencing localized musculoskeletal pain. To date there has been no evidence-based guidance generated to evaluate the efficacy of Multiprofen-CC™ in osteoarthritis patients. This study will test, in patients with end-stage knee osteoarthritis undergoing total knee arthroplasty, if the use of topical Multiprofen-CC™ in addition to standard of care pain management is more effective in controlling knee pain and reducing opioid use compared to placebo plus standard care alone.

DETAILED DESCRIPTION:
Total knee replacement, also known as total knee arthroplasty (TKA), is a surgical procedure aimed at alleviating pain and improving joint function in individuals with severe knee joint damage, often caused by conditions like osteoarthritis (OA) While TKAs generally yield positive results, a significant amount of patients express dissatisfaction with their outcomes, with some continuing to experience persistent pain after surgery. Opioids are very commonly prescribed for postsurgical pan, but they can cause a host of unwanted side effects. Orthopaedic surgeons prescribe opioids more frequently than in any other surgical speciality. This is a rising concern to the healthcare system as it may promote the development of opioid use disorder. There is a need for alternative therapies to opioid prescribing in patients having knee surgery to reduce the extensive health risks associated with opioid medications.

Multiprofen-CC™ is a multimodal topical cream including ingredients ketoprofen (10%), baclofen (5%), amitriptyline (2%), and lidocaine (5%). Healthcare professionals have the option to prescribe it to patients who are encountering localized musculoskeletal pain. To date there has been no evidence-based guidance generated to evaluate the efficacy of Multiprofen-CC™ in OA patients although there is compelling evidence that its medicinal ingredients are effective in pain relief.

The aim of the proposed study is to determine if, in patients with end-stage knee OA undergoing TKA, the use of topical Multiprofen-CC™ in addition to standard of care pain management is more effective in reducing acute post-operative pain during a 6 week follow-up period. Secondary objectives include determining the effects of Multiprofen-CC™ compared to placebo on opioid use, satisfaction with pain management, and we will also identify adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+)
* Undergoing Primary Elective TKA
* Provide informed consent

Exclusion Criteria:

* Administration of any investigational drug in the period of 0 to 45 days before entry into the study
* Pregnancy
* Actively breastfeeding
* Unable to provide informed consent (e.g. cognitive disability)
* Unable or unwilling to follow study protocol (e.g. unwilling to apply the topical treatments as instructed)
* Have a known allergy to ketoprofen, other NSAIDs, baclofen, amitriptyline, or lidocaine, any of the study drugs or their ingredients
* Have a history of substance abuse
* Use daily opioids (other than short acting codeine) for a chronic pain condition other than knee OA
* Are undergoing a revision TKA or are scheduled for a simultaneous bilateral TKA
* Any other condition which, in the opinion of the investigators, is likely to interfere with the successful collection of the measures required for the study
* Diagnosis of uncontrolled hypertension
* Diagnosis of active peptic ulcer disease
* A history of chronic (> 3 months) anticoagulant usage
* History of impaired kidney or liver function
* Have open wounds/cuts and/or skin conditions on the knee area, other than the surgical incision
* Body Mass Index (BMI) > 50kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain | 1, 2, 3, 4, 5, and 6 weeks postop
  Daily pain score on 0-10 numeric rating scale from post-op day 1 up to 6-weeks postop.

SECONDARY OUTCOMES:
Time to opioid cessation | 6 weeks postop
  Time to opioid cessation
Satisfaction with Pain Management | 6 weeks postop
  Satisfaction with pain management measured on a 0-10 numeric rating scale (NRS; higher score is better)
Safety - Adverse events | up to 6 weeks postop
  Serious and non-serious adverse events
Cumulative opioid use measured in Morphine Equivalent Dose (MED) | up to 6 weeks postop
  Cumulative opioid use up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Valente, MD, MMgt, FRCSC, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Oakville Trafalgar Memorial Hospital, Oakville, Ontario

IPD SHARING:
Plan to Share IPD: Undecided